CLINICAL TRIAL: NCT02210949
Title: Pre-operative Treatment With Erythropoietin and Iron Supplement for Prevention of Perioperative Blood Transfusion in Cardiac Surgery
Brief Title: Pre-operative Treatment With Erythropoietin and Iron Supplement in Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, AHM van Straten, MD, PhD, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPICSCZE14
Record Dates: First submitted 2014-06-23; First posted 2014-08-07 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Anemia, Iron-Deficiency
Keywords: Blood transfusion; Erythropoietin; Iron suppletion
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Epoetin Alfa; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythropoietin Iron (Other): Erythropoietin and iron:
  Administration of Erythropoietin (600 IU/kg (14.4 g/L)) twice weekly for three weeks .
  Administration of Iron (Ferinject (iron(III)carboxymaltose)) intravenously 1000 mg once.
  Interventions: Drug: Erythropoietin subcutaneously and Iron intravenously

INTERVENTIONS:
Drug: Erythropoietin subcutaneously and Iron intravenously — Administration of Erythropoietin subcutaneously and administration of iron intravenously
  Other Names: Eprex; Ferinject

SUMMARY:
Pre-treatment of patients with erythropoietin subcutaneously and iron supplement intravenously, in order to create a clinical pathway to minimize transfusion of red blood cells in a selected group of cardiac patients with an increased risk for blood transfusions in our cardiac surgery program.

DETAILED DESCRIPTION:
Blood transfusion is identified as an independent predictor of early mortality after Coronary artery bypass grafting operations In addition, female gender, lower body surface area (BSA), low preoperative Hemoglobin (Hb), previous cardiac surgery, emergency operation and low preoperative creatinin clearance were found to be independent risk factors for receiving Red Blood Cells (RBC) units.

We create a clinical pathway to reduce transfusion of red blood cells by pretreating patients with erythropoietin and iron to determine the reduction of number of patients who receive blood transfusion perioperatively. Also we want to investigate the decrease in the mean number of RBC units received per patient in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing isolated Coronary Artery Bypass Grafting operation or Aortic Valve Repair (AVR).
2. Preoperative Hb < 7 mmol/l.

Exclusion Criteria:

1. Off pump surgery.
2. Combination surgery.
3. Re-operation.
4. Emergency operation.
5. Patients with bleeding disturbances; e.g, hemophilia and patients with chronic liver disease.
6. Concomitant use of cyclosporine prior to, during or following surgery.
7. Female patients who are pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The number of patients who receive RBC transfusion perioperatively | 1 day
  To determine the reduction of the number of patients receiving blood transfusion the pre-treated group with erythropoietin and iron supplement compared to the control patients.
The number of patients who receive RBC transfusion perioperatively | 3 days
  To determine the reduction of the number of patients receiving blood transfusion the pre-treated group with erythropoietin and iron supplement compared to the control patients.
The number of patients who receive RBC transfusion perioperatively | 30 days
  To determine the reduction of the number of patients receiving blood transfusion the pre-treated group with erythropoietin and iron supplement compared to the control patients.

SECONDARY OUTCOMES:
To determine the degree of reduction in the mean number of RBC unit transfusions per patient. | 30 days
  In order to determine the degree of reduction in the mean number of RBC unit transfusions per patient. We count the units we need to give compared to the control group according to standard accepted postoperative levels Hb in our Hospital.

OTHER OUTCOMES:
Other general non specific outcome data after cardiac surgery | 30 days
  Moreover, early mortality and morbidity (postoperative blood loss, presence of myocardial infarction, Cerebral vascular accident (CVA), renal function disturbances) are always collected in the computerized database of the department of Cardiothoracic Surgery. These parameters will be used in the present study as well.

CONTACTS AND LOCATIONS:
Overall Officials: Marius C Haanschoten, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven the Netherlands
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] van Straten AH, Kats S, Bekker MW, Verstappen F, ter Woorst JF, van Zundert AJ, Soliman Hamad MA. Risk factors for red blood cell transfusion after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2010 Jun;24(3):413-7. doi: 10.1053/j.jvca.2010.01.001. Epub 2010 Mar 15. PMID 20231104
- [Background] Alghamdi AA, Albanna MJ, Guru V, Brister SJ. Does the use of erythropoietin reduce the risk of exposure to allogeneic blood transfusion in cardiac surgery? A systematic review and meta-analysis. J Card Surg. 2006 May-Jun;21(3):320-6. doi: 10.1111/j.1540-8191.2006.00241.x. PMID 16684074
- [Background] van Straten AH, Bekker MW, Soliman Hamad MA, van Zundert AA, Martens EJ, Schonberger JP, de Wolf AM. Transfusion of red blood cells: the impact on short-term and long-term survival after coronary artery bypass grafting, a ten-year follow-up. Interact Cardiovasc Thorac Surg. 2010 Jan;10(1):37-42. doi: 10.1510/icvts.2009.214551. Epub 2009 Oct 8. PMID 19815567
- [Background] Fox A. Recombinant human erythropoeitin: efficacy and safety considerations for maximizing blood conservation in cardiac surgery. Anesthesiology. 2011 Nov;115(5):912-4. doi: 10.1097/ALN.0b013e318231fd85. No abstract available. PMID 22027621